CLINICAL TRIAL: NCT01103921
Title: Effects of 2-weeks Fructose & HFCS Consumption on Dyslipidemia & Insulin Resistance
Brief Title: The Metabolic Effects of Consuming Sugar-Sweetened Beverages for Two Weeks
Acronym: DRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 200715772; R01HL091333 (NIH); R01HL107256 (NIH)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Dyslipidemia
Keywords: sugar; fructose; glucose; HFCS; metabolism
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Dyslipidemias | interventions — Glucose; Sugars; Fructose; High Fructose Corn Syrup; Aspartame

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Glucose (Other)
  Interventions: Other: Glucose
- Fructose (Other)
  Interventions: Other: Fructose
- High-Fructose Corn Syrup (Other)
  Interventions: Other: High-Fructose Corn Syrup
- Aspartame (Other): No sugar
  Interventions: Other: No sugar (Aspartame)

INTERVENTIONS:
Other: Glucose — 25% dose at 2-week intervention assigned to subjects.
  Other Names: Sugar
  Arms: Glucose
Other: Fructose — 25%, 17.5%, or 10% dose at 2-week intervention assigned to subjects.
  Other Names: Sugar
  Arms: Fructose
Other: High-Fructose Corn Syrup — 25%, 17.5%, or 10% dose at 2-week intervention assigned to subjects.
  Other Names: HFCS
  Arms: High-Fructose Corn Syrup
Other: No sugar (Aspartame) — 0% dose at 2-week intervention assigned to subjects.
  Other Names: Non-caloric sweetener
  Arms: Aspartame

SUMMARY:
The purpose of this study is to examine the effects of consumption of sugar-sweetened beverages on blood triglycerides and cholesterol, cholesterol concentrations, and the body's sensitivity to insulin.

DETAILED DESCRIPTION:
The study is designed as a prospective, blinded diet intervention study during which the participants consume either fructose- or HFCS-sweetened beverages (providing 10%, 17.5% or 25% of energy) with meals. In addition, there will be two control groups, with one group consuming 0% sugar beverages sweetened with sucralose and the other consuming glucose-sweetened beverages at 25% of energy requirement. Experimental procedures, including 24-hour serial blood sampling, post-heparin infusions, gluteal biopsies, Magnetic Resonance Imaging of the liver and the abdomen, and Oral Glucose Tolerance and Disposal Tests, are performed during baseline and at the end of a 2-week intervention period at the UC Davis Clinical and Translational Science Center (CTSC) Clinical Research Center (CCRC). During the inpatient periods, subjects are served energy balanced diets. The diets provide 15% of energy as protein, 30% as fat, and 55% as carbohydrate. During baseline testing, the carbohydrate content consists primarily of complex carbohydrate (>97%). During intervention the 55% carbohydrate will consist of 10% sugar/45% complex, 17.5% sugar/37.5% complex, or 25% sugar/30% complex depending on the diet group to which the subject is assigned. During the outpatient intervention periods, the subjects reside at home and are provided with fructose- or HFCS -sweetened beverages that are consumed with each meal along with a self-selected ad libitum (usual) diet.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18-35
* Self report of stable body weight during the past six months

Exclusion Criteria:

* Diabetes Mellitus
* Evidence of liver disorder
* Evidence of kidney disorder
* Evidence of thyroid disorder
* Systolic blood pressure consistently over 160mmHg or diastolic blood pressure over 900mmHg
* Triglycerides > 400mg/dl
* LDL-C > 240mg/dl
* Hemoglobin < 8.5 g/dl
* Current, prior (within 2 months), or anticipated use of any hypolipidemic or anti-diabetic agents
* Use of Selective Serotonin Reuptake Inhibitors and anti-hypertensive medications
* Any other condition that, in the opinion of the investigators, would put subject at risk
* Strenuous exerciser
* Pregnant or lactating women
* Smoker
* Diet exclusions: food allergies, special dietary restrictions, habitual ingest of >2 alcoholic beverages/day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2008-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
24-hour triglyceride area under the curve | Baseline and 2-week intervention
  32 serial blood samples are collected over a 24 hour period.

SECONDARY OUTCOMES:
Insulin sensitivity index | Baseline and 2-week intervention
  Insulin sensitivity is assessed using the deuterated glucose disposal method.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Havel, D.V.M, Principal Investigator — University of California, Davis; Kimber L Stanhope, Ph.D, R.D., Study Director — University of California, Davis
Locations (1):
- Clinical Research Center, Sacramento, California, United States

REFERENCES:
- [Derived] Sigala DM, Hieronimus B, Medici V, Lee V, Nunez MV, Bremer AA, Cox CL, Price CA, Benyam Y, Chaudhari AJ, Abdelhafez Y, McGahan JP, Goran MI, Sirlin CB, Pacini G, Tura A, Keim NL, Havel PJ, Stanhope KL. Consuming Sucrose- or HFCS-sweetened Beverages Increases Hepatic Lipid and Decreases Insulin Sensitivity in Adults. J Clin Endocrinol Metab. 2021 Oct 21;106(11):3248-3264. doi: 10.1210/clinem/dgab508. PMID 34265055
- [Derived] Hieronimus B, Medici V, Bremer AA, Lee V, Nunez MV, Sigala DM, Keim NL, Havel PJ, Stanhope KL. Synergistic effects of fructose and glucose on lipoprotein risk factors for cardiovascular disease in young adults. Metabolism. 2020 Nov;112:154356. doi: 10.1016/j.metabol.2020.154356. Epub 2020 Sep 9. PMID 32916151
- [Derived] Stanhope KL, Medici V, Bremer AA, Lee V, Lam HD, Nunez MV, Chen GX, Keim NL, Havel PJ. A dose-response study of consuming high-fructose corn syrup-sweetened beverages on lipid/lipoprotein risk factors for cardiovascular disease in young adults. Am J Clin Nutr. 2015 Jun;101(6):1144-54. doi: 10.3945/ajcn.114.100461. Epub 2015 Apr 22. PMID 25904601
- [Derived] Tryon MS, Stanhope KL, Epel ES, Mason AE, Brown R, Medici V, Havel PJ, Laugero KD. Excessive Sugar Consumption May Be a Difficult Habit to Break: A View From the Brain and Body. J Clin Endocrinol Metab. 2015 Jun;100(6):2239-47. doi: 10.1210/jc.2014-4353. Epub 2015 Apr 16. PMID 25879513